CLINICAL TRIAL: NCT05185115
Title: Efficacy of Nasal Oxygen Therapy to Reduce Postoperative Complications in Ankle Trauma Surgery in At-risk Patients: a Randomized Pilot Study
Acronym: TOP-ANK
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC21_0129
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (A) (Experimental): Patients treated with 3 liters per minute oxygen delivered via nasal cannula duration hospitalization
  Interventions: Drug: Oxygen
- Control group (B) (Other): No oxygen therapy during hospitalization
  Interventions: Other: no oxygen therapy

INTERVENTIONS:
Drug: Oxygen — administration of oxygen at a flow rate of 3 liters per minute, via nasal cannula throughout the hospitalization.
  Other Names: O2
  Arms: Intervention group (A)
Other: no oxygen therapy — No oxygen therapy during hospitalization
  Arms: Control group (B)

SUMMARY:
Ankle fractures are one of the most common surgeries in the world. After this kind of surgery, complications can occur, related to the scar or an infection. These complications are more frequent in "high-risk" patients. Nasal oxygen therapy is currently used in order to reduce these complications. However, no study proved its efficiency yet. In a cohort of 200 patients, one group will receive oxygen therapy during hospitalization, while the other will not. Complication rates will be observed up to 6 months after the operation

DETAILED DESCRIPTION:
Prospective, single-center, comparative and randomized study based on a cohort of 200 patients with an ankle fracture. The patients will be assigned to one of the following group: with or without oxygen therapy. Patients in the experimental group will receive the oxygen just before the operation, and during the hospitalization. The rest of the care is the same for the 2 groups. Comparison of complication rate, of quality of healing, rate of revision surgery, delay in bone healing, rate of pseudoarthrosis, and ankle pain will be done between the 2 groups during a postoperative period of 6 months. A cost-utility analysis will also be realized. In a subgroup of 40 patients, additional transcutaneous oxygen pressure measurements will be performed to compare the evolution of tissue oxygenation between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with an ankle joint injury with surgical indication
* Patient with at least one risk factor for scar complication such as comorbidity(ies) (diabetes, smoking, peripheral neuropathy, obstructive arterial disease of the lower limbs, microangiopathy, treatment influencing healing (chemotherapy, corticosteroids...)) and/or complex fracture
* Patient affiliated to a social security system
* Patient having signed an informed consent

Exclusion Criteria:

* Patient with chronic respiratory insufficiency
* Patient with sleep apnea with equipment
* Patient under long term oxygen therapy
* Patient with a bilateral ankle fracture
* Polytrauma patients
* Pregnant or breastfeeding women or those refusing effective contraception
* Patient deprived of liberty or under legal protection (guardianship or curatorship)
* Patient unable to follow the protocol, as judged by the investigator
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-09 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Cutaneous and infectious complications | 6 months
  Post-surgery ankle complications including skin damage (ecchymosis, phlyctena), necrosis, superficial and deep infection and scar disunion

SECONDARY OUTCOMES:
Observer Scar Assessment Scale (OSAS questionnaire) | 3 weeks after surgery
  The OSAS grid is used to evaluate the tolerance and scar quality obtained by the operator. It is based on an evaluation of the healing process thanks to 7 questions whose answers are rated according to an increasing scale from 1 to 10 (1 corresponding to the best result and 10 the worst). The result will lead to a score of 7 to 70 points
Observer Scar Assessment Scale (OSAS questionnaire) | 6 weeks after surgery
  The OSAS grid is used to evaluate the tolerance and scar quality obtained by the operator. It is based on an evaluation of the healing process thanks to 7 questions whose answers are rated according to an increasing scale from 1 to 10 (1 corresponding to the best result and 10 the worst). The result will lead to a score of 7 to 70 points
Observer Scar Assessment Scale (OSAS questionnaire) | 12 weeks after surgery
  The OSAS grid is used to evaluate the tolerance and scar quality obtained by the operator. It is based on an evaluation of the healing process thanks to 7 questions whose answers are rated according to an increasing scale from 1 to 10 (1 corresponding to the best result and 10 the worst). The result will lead to a score of 7 to 70 points
Revision surgery | 6 months after surgery
Pseudoarthrosis Complication | 24 weeks after surgery
  Presence of delayed healing on radiograph at S24
Visual Analogue Scale (VAS) to evaluate ankle pain | preoperatively
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Visual Analogue Scale (VAS) to evaluate ankle pain | 24 hours after surgery
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Visual Analogue Scale (VAS) to evaluate ankle pain | 48 hours after surgery
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Visual Analogue Scale (VAS) to evaluate ankle pain | 3 weeks after surgery
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Visual Analogue Scale (VAS) to evaluate ankle pain | 6 weeks after surgery
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Visual Analogue Scale (VAS) to evaluate ankle pain | 12 weeks after surgery
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Visual Analogue Scale (VAS) to evaluate ankle pain | 24 weeks after surgery
  The VAS measures the intensity of pain on a scale from 0 to 10 (0= no pain ans 10 = worst pain)
Transcutaneous oxygen pressure measurements (TcPO2) | before the initiation of oxygen therapy preoperatively
  The Measurement of TcPO2 will be performed in a subgroup of 40 patients (20 patients in each group)
Transcutaneous oxygen pressure measurements (TcPO2) | 48hours after surgery
  The Measurement of TcPO2 will be performed in a subgroup of 40 patients (20 patients in each group)
Transcutaneous oxygen pressure measurements (TcPO2) | 3 weeks after surgery
  The Measurement of TcPO2 will be performed in a subgroup of 40 patients (20 patients in each group)
EuroQol 5-Dimension (EQ-5D) self-questionnaire | pre-operatively
  This quality of life questionnaire is completed in order to realize a cost-utility analysis (cost per QALY)
EuroQol 5-Dimension (EQ-5D) self-questionnaire | 48 hours after surgery
  This quality of life questionnaire is completed in order to realize a cost-utility analysis (cost per QALY)
EuroQol 5-Dimension (EQ-5D) self-questionnaire | 3 weeks after surgery
  This quality of life questionnaire is completed in order to realize a cost-utility analysis (cost per QALY)
EuroQol 5-Dimension (EQ-5D) self-questionnaire | 6 weeks after surgery
  This quality of life questionnaire is completed in order to realize a cost-utility analysis (cost per QALY)
EuroQol 5-Dimension (EQ-5D) self-questionnaire | 12 weeks after surgery
  This quality of life questionnaire is completed in order to realize a cost-utility analysis (cost per QALY)
EuroQol 5-Dimension (EQ-5D) self-questionnaire | 24 weeks after surgery
  This quality of life questionnaire is completed in order to realize a cost-utility analysis (cost per QALY)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Gadbed, Nantes, France, France

IPD SHARING:
Plan to Share IPD: No